CLINICAL TRIAL: NCT06411054
Title: The Efficacy of Acupuncture-type Transcutaneous Electrical Nerve Stimulation as an Adjunct Analgesic in Reducing Pain During Ultrasound-guided Manual Vacuum Aspiration: A Prospective, Single- Blinded Two-arm Randomized Controlled Trial.
Brief Title: The Efficacy of Acu-TENS as an Adjunct Analgesic During USG-MVA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Chung Pui Wah Jacqueline, Associate Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CRE-2023.578
Record Dates: First submitted 2024-04-29; First posted 2024-05-13 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Pain, Acute
Keywords: Manual vacuum aspiration; Ultrasound-guided; Acupuncture transcutaneous electrical nerve stimulation; Alternative medicine; Randomized controlled trial
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Au-TENS group (Experimental): Women will receive acu-TENS from 15 minutes before USG-MVA to 15 minutes after USG-MVA.
  Interventions: Device: Acu-TENS
- Sham acu-TENS group (Sham Comparator): Women will receive sham acu-TENS from 15 minutes before USG-MVA to 15 minutes after USG-MVA. In the sham acu-TENS, TENS pads will be placed on the same acupoints, connected to the machine, but without electric current.
  Interventions: Device: Sham acu-TENS

INTERVENTIONS:
Device: Acu-TENS — After cleaning the acupoints with alcohol, electrode pads (HC-ROUND-32 2.0) will be placed on the acupoints SP6, ST36, LI4, LR3, according to the locations described in the Standard International Acupuncture Nomenclature. The electrode pads will be connected to a TENS machine (MTRP-00003), in which ipsilateral LI4 and SP36, SP6 and LR3 serve a pair. A pulse rate of 120 Hz, current of 4-12mA, and pulse width of 300µS will be delivered continually for 45 minutes (i.e. from 15 minutes before starting the MVA to 15 minutes after the procedure has completed).
  Arms: Au-TENS group
Device: Sham acu-TENS — After cleaning the acupoints with alcohol, electrode pads (HC-ROUND-32 2.0) will be placed on the acupoints SP6, ST36, LI4, LR3, according to the locations described in the Standard International Acupuncture Nomenclature. The electrode pads will be connected to a TENS machine (MTRP-00003), in which ipsilateral LI4 and SP36, SP6 and LR3 serve a pair.
  In the sham acu-TENS, TENS pads will be placed on the same acupoints, connected to the machine, but without electric current. The pads will be stuck on the acupoints for 45 minutes (i.e. from 15 minutes before starting the MVA to 15 minutes after the procedure has completed).
  Arms: Sham acu-TENS group

SUMMARY:
Objectives: To prospectively evaluate the potential of acu-TENS to reduce the pain experienced by women undergoing ultrasound-guided manual vacuum aspiration (USG-MVA) and evaluate its safety profile.

Hypothesis to be tested: Does the use of acu-TENS reduce pain in women undergoing USG-MVA?

Design and subjects: A prospective randomized control trial will be carried out at the Department of Obstetrics and Gynaecology of the Prince of Wales Hospital. Women undergoing USG-MVA for the treatment of early pregnancy loss before 12 weeks of gestation will be randomized to receive acu-TENS (intervention group) or sham acu-TENS (control group) for pain control during USG-MVA. We will recruit 54 participants in each of the two arms, so a total of 108 patients will be recruited.

Study instruments: USG-MVA will be performed using a 60ml charged syringe (MedGyn Aspiration Kit) with a flexible curette attached to it. Transabdominal ultrasound during the MVA procedure will be performed using Mindray DC-80A Diagnostic Ultrasound System. Acu-TENS will be performed using MTR+ Myolito Multifunctional Stimulator (MTRP-00003).

Main outcome measures: Primary outcome includes pain scores before, during and after USG-MVA. Secondary outcomes include (1) stress levels measured by heart rate, heart rate variability, blood pressure, State Trait Anxiety Inventory (STAI), and salivary cortisol; (2) anxiety level; (3) Surgeon's assessment on the patient co-operation score and patient intraoperative pain, (4) Client Satisfaction Questionnaire (CSQ8) and satisfaction score, and (5) any adverse events of acu-TENS.

Data analysis: Data analysis will be performed using the Statistical Packages of Social Sciences for Windows (SPSS, Inc).

Expected results: We expect that acu-TENS will result in at least a 35% reduction in pain experienced by women undergoing USG-MVA.

DETAILED DESCRIPTION:
Randomization process and blinding of clinician For those who consented to the study, they will be randomly assigned preoperatively to receive "acu-TENS" or "sham acu-TENS" according to a computer-generated random number series by an independent research nurse who is not in our team in a 1:1 ratio. Prior to the onset of the study, sequentially numbered (written on top) non-opaque envelopes containing treatment modality, (i) intervention group (Group A): acu-TENS in USG-MVA (ii) controlled group (Group B): sham acu-TENS in USG-MVA will be also prepared by an independent research nurse. On opening the envelope, the study nurse will record the envelope number and the randomization group assigned in patient recruitment password protected electronic file. The assigned envelope number will then be documented in a second electronic password protected file which will be used to document procedure details, patients' details, procedure outcome and investigation assessments.

The Firstbeat Body-guard 3 device to measure HRV will be applied 1 hour before the procedure and will remain in place for 1 hour after the procedure.

15 minutes before MVA, after the clinician has applied the TENS pads on specific acupoints, and connected the pads to the TENS machine, the study nurse will be responsible to (i) intervention group (Group A): turn on the TENS machine or (ii) controlled group (Group B): pretend to turn on the TENS machine. 15 minutes after MVA, the study nurse will (i) intervention group (Group A): turn off the TENS machine or (ii) controlled group (Group B): pretend to turn off the TENS machine. After that, the clinician will disconnect the wires and remove the pads. Hence, the clinician will be blinded throughout the process.

The study nurse will not be present during the operative procedure, nor will she be involved in the any investigations. Moreover, another team of gynaecologist and nursing staff will help with the follow-up phone calls to avoid performance and measurement biases and the problem of automatic unblinding.

USG-MVA procedure All women will be asked to fill in the STAI questionnaire before they come to hospital. Once admitted, all women will be given 400µg of misoprostol orally for cervical priming, 2-3 hours before the procedure. 500mg of naproxen will be given 60 min before the procedure. Paracetamol or codeine will be used as an alternative to naproxen in case of allergy.

The USG-MVA procedure will be carried out by doctors with similar surgical experience who have carried out at least 25 USG-MVA procedures independently. The USG-MVA will be carried out using a 60-ml charged syringe (MedGyn Aspiration Kit IV, 022511) (Addison, IL, USA) with a flexible curette (size 4-7 mm, subject to the doctor's discretion) attached to it. Paracervical block will be carried out using a 23-gauge dental needle syringe to inject 5 ml of 2% lidocaine into a depth of 0.5 cm at the cervical-vaginal juncture at 4, 5, 7 and 8 o'clock position to reach the uterosacral ligaments. A tenaculum will be used to hold the cervix if necessary. Voluson E730 Expert USG system will be used for transabdominal USG during MVA. During the procedure, 5-ml of local lidocaine gel will be applied to the cervical canal and over the end of the MVA catheter tip during the insertion. A research assistant will help the patient with filling in an intra-procedure VAS questionnaire.

The USG-MVA procedure will be stopped as soon as the operating clinician is satisfied that the uterine cavity is empty. Products of conception will be sent for histological evaluation and cytogenetic analysis if clinically indicated. Postoperative complications, including significant bleeding requiring blood transfusion, uterine perforation and infection and side-effects such as nausea, vomiting, dizziness, drowsiness, shortness of breath and dry mouth or eyes from the medication and their severity will be documented.

Acu-TENS treatment and Sham acu-TENS treatment All acu-TENS and sham acu-TENS treatments will be performed on site in the same manner by a clinician who follows a standard approach to describe the intervention to participants.

After cleaning the acupoints with alcohol, electrode pads (HC-ROUND-32 2.0) will be placed on the acupoints SP6, ST36, LI4, LR3, according to the locations described in the Standard International Acupuncture Nomenclature. The electrode pads will be connected to a TENS machine (MTR+ Myolito Multifunctional Stimulator MTRP-00003), in which ipsilateral LI4 and SP36, SP6 and LR3 serve a pair. A pulse rate of 120 Hz, current of 4-12mA, and pulse width of 300µS will be delivered continually for 45 minutes (i.e. from 15 minutes before starting the MVA to 15 minutes after the procedure has completed).

In the sham acu-TENS group, TENS pads will be placed on the same acupoints, connected to the machine, but without electric current.

Measurement of Pain Individual pain scores, measured by the visual analog scale (VAS), is recorded before taking misoprostol, right before the surgery, during (during cannula insertion, and for every suction), and after USG-MVA (0 min, 15 min, 30 min, and 1-hour post-MVA). Women will be asked to move the cursor along the VAS ruler, which does not have markings other than '0' and '10', to indicate her pain level at different time intervals. With a change of more than or equal to 10 for the 100 mm VAS, the analgesic intervention is clinical important.

To validate the VAS pain score rated by patients, surgeons will rate the patient compliance index and patient pain score. For the patient compliance index, it is a 5-point Likert scale rated from 1 (fully co-operation) to 5 (no co-operation, procedure abandoned).For the patient pain score, it is a 5-point Likert scale rated from 0 (patient did not show any sign of pain) to 4 (patient did not let the procedure continue which was demonstrated by verbal or bodily expression).

Measurement of stress

1. Blood pressure will be recorded before taking misoprostol, right before the surgery, during (during cannula insertion, and for every suction), and after USG-MVA (0 min, 15 min, 30 min, and 1-hour post-MVA).
2. Heart rate and HRV one hour before USG-MVA to one hour after USG-MVA will be measured using Firstbeat Bodyguard 3 devices. Studies have shown that in acute pain, with ascending nociception, segmental spinal reflexes are recruited to activate the sympathetic system, resulting in increased peripheral resistance, heart rate, and stroke volume). HRV is a non-invasive measurement of the variation in time between consecutive heartbeats which provides information about the balance between the sympathetic (fight-or-flight) and parasympathetic (rest-and-digest) branches of the autonomic nervous system. Under high stress, amygdala activation initiates the hypothalamic-pituitary-adrenal axis (HPA axis) response and parasympathetic withdrawal. This enhanced stress load is expressed as decreased cardiac vagal activity. HRV has also been found to be a useful in evaluating pain response and can potentially overcome some of the challenges of quantifying pain.
3. Saliva will be collected for cortisol analysis before, immediately after, and 15 minutes after MVA. Cortisol is a stress hormone. We test the cortisol level in saliva instead of blood to avoid the stress brought by blood drawing which will result in elevated cortisol levels. Studies indicate elevated saliva cortisol levels in pain, for example, fibromyalgia and myofascial pain. Vice versa, when pain is relieved, saliva cortisol level will decrease. For example, pain is relieved by dance and yoga in functional abdominal pain disorders.
4. Participants will be asked to fill in the STAI questionnaire before and after USG-MVA. STAI is a 40-items scale which used 4-point Likert scale ranged from almost never to almost always. The higher scoring indicates greater level of anxiety. It consists of two parts, the S-AD questionnaire for stress level and the T-AI questionnaire for traits. The validated Chinese version of STAI was used to measure the changing psychological status before and after USG-guided MVA, with a score ranging from 20 to 80. Participants will be asked to fill in both parts when they arrived at the hospital. This can give a better baseline anxiety index. A stress state may affect the pain level. Hence, after the USG-MVA procedure, the S-AD questionnaire will be done again.

Measurement of anxiety Participants will be asked to rate the VAS-anxiety before and after the USG-MVA procedure.

Measurement of patient satisfaction Participants will be asked to complete a client satisfaction questionnaire (CSQ8) after USG-MVA. CSQ8 contains eight items including the concern of quality of service, kind of service, outcome of service, extent in meeting their need, recommendation to friend, amount of help, effectiveness in dealing the problem, overall satisfaction and willingness to use the service again. It is rated by four-point Likert scale, which scores ranged from 8 to 32. The higher scores indicate greater satisfaction with the service or treatment. Participants will also be asked to rate their satisfaction on the MVA service from 0 score (lowest satisfaction) to 100 score (highest satisfaction) by a 100mm scale.

Recording the safety profile and potential benefits Follow-up phone calls will be made 1 month after the procedure to ask for possible side effects. Any serious adverse effects will be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 or above;
2. Patient diagnosed with first-trimester miscarriage, who is eligible for USG-MVA;
3. Patient diagnosed with incomplete miscarriage after medical treatment;
4. Willing to be randomized to receive acupuncture.

Exclusion criteria

a. Patient not eligible for USG-MVA i. Miscarriage > 12 weeks of gestation; or ii. Pregnancy of unknown origin; or iii. Known narrowing of the cervical canal; or iv. Multiple uterine fibroids; or v. Congenital uterine anomalies; or vi. Active pelvic infection; or vii. Bleeding disorder; or viii. Inability to tolerate pelvic examination; or ix. History of allergy to misoprostol

b. Patient not eligible for acu-TENS i. Poor skin integrity at the acupuncture site, such as open wound, infections, unknown mass, bleeding tendency; or ii. Allergic to external alcohol; or iii. Emotionally unstable or tend to restlessness (to avoid tear-off of pads).

c. Patient refusal

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 108 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
VAS pain score | Before taking misoprostol, right before the surgery, during (during cannula insertion, and for every suction), and after USG-MVA (0 minutes, 15 minutes, 30 minutes, and 1-hour post-USG-MVA)
  Women will be asked to move the cursor along the VAS ruler, which does not have markings other than '0' and '10', to indicate her pain level at different time intervals. With a change of more than or equal to 10 for the 100 mm VAS, the analgesic intervention is clinical important (Myles et al., 2017).

SECONDARY OUTCOMES:
Stress level measured by STAI questionnaire | 2 hours before and 1 hour after USG-MVA
  STAI is a 40-items scale which used 4 point Likert scale ranged from almost never to almost always. It consists of two parts, the S-AD questionnaire for stress level and the T-AI questionnaire for traits. The validated Chinese version of STAI was used to measure the changing psychological status before and after USG-guided MVA, with a score ranging from 20 to 80.
Stress level measured by saliva cortisol | 2 hours before, right after, and 30 minutes after USG-MVA
  We test the cortisol level in saliva instead of blood to avoid the stress brought by blood drawing which will result in elevated cortisol levels. Studies indicate elevated saliva cortisol levels in pain, for example, chronic widespread pain or fibromyalgia(Begum et al., 2022), and myofascial pain(Nadendla et al., 2014). Vice versa, when pain is relieved, saliva cortisol level will decrease. For example, pain is relieved by dance and yoga in functional abdominal pain disorders(Areskoug Sandberg et al., 2022).
VAS Anxiety Score | Before taking misoprostol, right before the surgery, during (during cannula insertion, and for every suction), and after USG-MVA (0 minutes, 15 minutes, 30 minutes, and 1-hour post-USG-MVA)
  Women will be asked to move the cursor along the VAS ruler, which does not have markings other than '0' and '10', to indicate her pain level at different time intervals.
Blood pressure | Before taking misoprostol, right before the surgery, during (during cannula insertion, and for every suction), and after USG-MVA (0 minutes, 15 minutes, 30 minutes, and 1-hour post-USG-MVA)
  Studies have shown that in acute pain, with ascending nociception, segmental spinal reflexes are recruited to activate the sympathetic system, resulting in increased peripheral resistance, heart rate, and stroke volume(Bruehl et al., 2010; Fagius et al., 1989; Saccò et al., 2013(Bruehl et al., 2002)).
Heart rate and heart rate variability | One hour before USG-MVA to one hour after USG-MVA
  Studies have shown that in acute pain, with ascending nociception, segmental spinal reflexes are recruited to activate the sympathetic system, resulting in increased peripheral resistance, heart rate, and stroke volume(Bruehl et al., 2010; Fagius et al., 1989; Saccò et al., 2013(Bruehl et al., 2002)).
Patient Satisfaction Score | One hour after USG-MVA
  Participants will also be asked to rate their satisfaction on the MVA service from 0 score (lowest satisfaction) to 100 score (highest satisfaction) by a 100mm scale.
Client satisfaction questionnaire (CSQ8) | One hour after USG-MVA
  CSQ8 contains eight items including the concern of quality of service, kind of service, outcome of service, extent in meeting their need, recommendation to friend, amount of help, effectiveness in dealing the problem, overall satisfaction and willingness to use the service again. It is rated by four-point Likert scale, which scores ranged from 8 to 32. The higher scores indicate greater satisfaction with the service or treatment.
Patient compliance index | Right after USG-MVA
  To validate the VAS pain score rated by patients, surgeons will rate the patient compliance index. It is a 5-point Likert scale rated from 1 (fully co-operation) to 5 (no co-operation, procedure abandoned).
Patient pain score | Right after USG-MVA
  To validate the VAS pain score rated by patients, surgeons will rate the patient pain score. It is a 5-point Likert scale rated from 0 (patient did not show any sign of pain) to 4 (patient did not let the procedure continue which was demonstrated by verbal or bodily expression).
Potential benefits | 1 year post USG-MVA
  Pregnancy outcomes, information collected by phone calls
Adverse events | 1 month post USG-MVA
  Information collected by phone calls

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong